CLINICAL TRIAL: NCT04069377
Title: Mechanical Versus Manual Chest Compression: A Retrospective Study in Out-of-hospital Cardiac Arrest
Brief Title: Mechanical Versus Manual Chest Compression
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Collaborators: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Alp Şener, Clinical Assistant Professor, Ankara City Hospital Bilkent
Other Study IDs: medybu154
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Cardiac Arrest; Cardiopulmonary Resuscitation
Keywords: Cardiopulmonary Resuscitation; Chest compression; Manuel; Mechanical
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Manuel chest compression: Manuel chest compressions will be handled by human efforts.
  Interventions: Other: Manuel chest compressions by human efforts
- Mechanical chest compression: In the study, chest compression in the mechanical cardiopulmonary resuscitation group was performed with the Lund University Cardiopulmonary Assist System (LUCAS) Chest Compression System (LUCAS 2).
  Interventions: Device: LUCAS™ 2 Chest Compression System

INTERVENTIONS:
Device: LUCAS™ 2 Chest Compression System — LUCAS is a portable device designed to rule out the problems encountered during manual chest compression, capable of performing standard and continuous chest compressions at a depth of 4-5 cm and at least 100 times per minute.
  Groups: Mechanical chest compression
Other: Manuel chest compressions by human efforts — In this way chest compressions will be handled by humans themselves.
  Groups: Manuel chest compression

SUMMARY:
In this study, the investigators compared mechanical and manual chest compressions in out-of-hospital cardiac arrest cases.

DETAILED DESCRIPTION:
In this study, the investigators retrospectively analyzed resuscitations performed over a 2-year period and compared manual and mechanical chest compressions in terms of return of spontaneous circulation, 30-day survival, and hospital discharge parameters.

ELIGIBILITY:
Inclusion Criteria:

Over 18 age Cardiac arrest cases Out-of-hospital arrest

Exclusion Criteria:

<18 age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The data of out-of-hospital cardiac arrest cases undergoing cardiopulmonary resuscitation in the emergency department were analyzed retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-04-15 (Actual)

PRIMARY OUTCOMES:
Rate of the mortality on the 30th day | 30 days
  Mortality from the admission to the 30th day
Rate of the return of spontaneous circulation | 5 minutes
  Return of spontaneous circulation at least 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, School of Medicine, Department of Emergency Medicine, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) with other researchers.

REFERENCES:
- [Background] Brodal Syversen K, Souvannasacd E, Renger R. Validating the LUCAS(R) mechanical chest compression fit specifications. Am J Emerg Med. 2019 Feb;37(2):371-373. doi: 10.1016/j.ajem.2018.06.069. Epub 2018 Jun 30. No abstract available. PMID 30686332
- [Background] Bonnes JL, Brouwer MA, Navarese EP, Verhaert DV, Verheugt FW, Smeets JL, de Boer MJ. Manual Cardiopulmonary Resuscitation Versus CPR Including a Mechanical Chest Compression Device in Out-of-Hospital Cardiac Arrest: A Comprehensive Meta-analysis From Randomized and Observational Studies. Ann Emerg Med. 2016 Mar;67(3):349-360.e3. doi: 10.1016/j.annemergmed.2015.09.023. Epub 2015 Nov 19. PMID 26607332
- [Background] Gates S, Quinn T, Deakin CD, Blair L, Couper K, Perkins GD. Mechanical chest compression for out of hospital cardiac arrest: Systematic review and meta-analysis. Resuscitation. 2015 Sep;94:91-7. doi: 10.1016/j.resuscitation.2015.07.002. Epub 2015 Jul 17. PMID 26190673